CLINICAL TRIAL: NCT06887647
Title: Physical Therapy for Montana Children With Neuromotor Disorders Using Hippotherapy and the Equine Environment
Brief Title: PT for Montana Children With NMD Using Hippotherapy and the Equine Environment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Montana (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-FY2024-330; P20GM103474 (NIH)
Record Dates: First submitted 2025-03-10; First posted 2025-03-20 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-03

CONDITIONS: Neuromotor Impairments
Keywords: physical therapy; hippotherapy; pediatric; motor function; participation; upper extremity function; equine environment; neurmotor disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Play-Based Physical Therapy (Active Comparator): Participants in the control group will receive 8 weeks of standard play-based PT, 2 x 1-hour sessions per week, for a total of 16 hours. The sessions will be implemented by a licensed PT.
  Interventions: Other: Standard Play-Based Physical Therapy
- Physical Therapy Using Hippotherapy and the Equine Environment (Experimental): Participants in the intervention group will receive 8 weeks of PT using hippotherapy and the equine environment, 2 x 1-hour sessions per week (16 hours total). Treatment will be provided by a licensed PT with the recommended training to incorporate hippotherapy and the equine environment into treatment (American Hippotherapy Association (AHA) Inc. Hippotherapy Treatment Principles Part I and II). Each therapist will work with an equine professional with PATH Intl. Therapeutic Riding Instructor Certification, to ensure that therapists adhere to industry standards for safety and handling of the equines.
  Interventions: Other: Physical Therapy Using Hippotherapy and the Equine Environment

INTERVENTIONS:
Other: Physical Therapy Using Hippotherapy and the Equine Environment — Subjects will be mounted on a horse for 15-30 minutes. Therapeutic activities will include movements like reaching, throwing, and bilateral coordination tasks in addition to assuming various positions on the horse during equine movement, per the tolerance of individual participants. Remaining treatment time will involve participation-based functional motor activities in the equine environment, such as feeding and grooming horses.
  Treatment will include the following active ingredients:
  1. Encourage use of both upper extremities during therapeutic activities.
  2. Design therapeutic activities with equines to guide practice of functional motor skills.
  3. Design therapeutic activities with the equines to practice participation (ie. activities involved in life situations).
  4. Utilize the presence of the equines to optimize patient mood and engagement in the therapeutic activities. (Design activities around patient strengths and preferences; use the equines as positive reinforcement)
  Arms: Physical Therapy Using Hippotherapy and the Equine Environment
Other: Standard Play-Based Physical Therapy — The treatment will focus on encouragement of functional play activities, such as reaching, throwing, and catching games. Treatment will incorporate the following active ingredients:
  1. Encourage use of both upper extremities during therapeutic activities.
  2. Design therapeutic activities using play and games to guide practice of functional motor skills.
  3. Design therapeutic activities with play and games to practice participation (ie. activities involved in life situations).
  4. Utilize play and games to optimize patient mood and engagement in the therapeutic activities. (Design activities around patient strengths and preferences; use play and games as positive reinforcement)
  Arms: Play-Based Physical Therapy

SUMMARY:
The goal of this pilot clinical trial is to determine if physical therapy incorporating horses can improve the motor skills of the arms in children 6-17 years old with neuromotor disorders (such as cerebral palsy, spinal muscular atrophy, or spina bifida) compared to standard play-based physical therapy. The main questions it aims to answer are:

1. Is the study protocol feasible and acceptable for participants, that investigators could apply them to a larger trial?
2. Do participants make improvements toward their goals for motor function, arm use, and participation in life situations following treatment, and is it different between the experimental and comparative intervention groups?
3. What are the physiological, behavioral, and emotional responses of children receiving physical therapy incorporating horses, versus those receiving standard physical therapy?

Researchers will compare the experimental group who receive physical therapy incorporating horses to the comparative intervention group who receive standard play-based physical therapy to see if there is a difference in outcomes.

Participants will complete a pre- and post-intervention assessment of their motor function and participation in life situations. Participants will receive physical therapy twice a week for 8 weeks for the intervention. In both groups, physiological, behavioral, and emotional responses to the interventions will be measured in 4 total sessions, 1 each at weeks 2, 4, 6, and 8.

DETAILED DESCRIPTION:
The long-term goal is to increase the variety of effective PT interventions for children with NMD, to achieve optimum outcomes for all. The investigators have already completed a pilot feasibility randomized-controlled trial (RCT) with waitlist control of an intervention targeting upper extremity function and participation in children with neuromotor disorders. The intervention protocol was feasible, but certain aspects of the RCT protocol needed to be revised. Aim 1 of this proposal evaluates the feasibility of these revisions by: 1) establishing an appropriate control condition, 2) evaluating replacement outcome measures for those that were not feasible; and 3) determining effects of a different treatment dosage on retention and attendance. Aim 2 will explore preliminary effects of the intervention on motor function and participation and Aim 3 will explore behavioral and physiological responses.

Aim 1: Evaluate the feasibility of the RCT protocol comparing an 8-week PT intervention using hippotherapy and the equine environment with a play-based PT control group targeting motor function and participation for children with NMD. Inestigators will track recruitment, retention, attendance, outcome measure completion, and reasons for absences and withdrawal. Investigators will assess fidelity and acceptability of the treatments for both groups. This will inform design of a large-scale RCT with full statistical power. Investigators hypothesize that they will recruit and randomize 24 participants with >80% retention, treatment attendance, and outcome measure completion in both groups; and both groups will meet >80% intervention fidelity and demonstrate acceptability.

Aim 2: Identify preliminary effects of an 8-week PT intervention using hippotherapy and the equine environment on motor function and participation compared to play-based PT for children with NMD. Investigators will measure motor function (BOT-3, ABILHANDKIDS), individual goal attainment (GAS), and participation (PEM-CY) before and after the 8-week treatment period for all participants and compare the average change score between the treatment and control groups. Investigators hypothesize that group average scores will improve from pre- to post-treatment for both groups, with a greater change in the treatment group compared to the control group.

Aim 3: Compare physiological, behavioral, and emotional responses in children with NMD during PT sessions incorporating equine interaction versus play-based PT. Investigators will calculate changes in high-frequency heart rate variability (HF-HRV) - the gold standard method of measuring parasympathetic nervous system activity - before, during, and after a treatment session. Investigators will measure levels of salivary oxytocin and cortisol before and after a treatment session. Investigators will assess engagement during treatment using behavioral coding and an observational rating scale. Enjoyment will be measured via patient report on a visual-analog scale following treatment. These measures will be collected during 4 treatment sessions (every 2 weeks) throughout the intervention. Investigators hypothesize that the intervention group will demonstrate an immediate increase in HF-HRV and salivary oxytocin, and a decrease in salivary cortisol after a single 60-minute session and sustained over the course of the 8-week intervention; participants will demonstrate sustained high engagement and enjoyment over the course of the intervention, and ratings of engagement and enjoyment will be greater than in the control condition; and physiological changes and behavioral ratings will be significantly positively correlated with the outcomes measured in Aim 2.

Background and Rationale There is a growing number of children with NMD across the United States. In rural areas like Montana, access and adherence to PT is especially challenging. Offering PT services in an equine environment can increase access to rural populations and provide PT in setting that might be more motivating and engaging for children, however there is a need to further evaluate its efficacy for improving important outcomes, like motor function and participation. The investigators began to address this need with a previous feasibility RCT which is linked in References. In Aim 1 investigators will implement changes identified to improve feasibility of the RCT protocol: 1) add additional screening to confirm that participants can complete all measures; 2) assess the feasibility of a play-based PT control condition; 3) test the reduced frequency of 2x/ week with a larger sample, and 4) replace the outcome measures that had low completion rates. Results from Aim 1 will inform the design of a large-scale clinical efficacy trial. In Aim 2, investigators will evaluate preliminary efficacy of the PT intervention using hippotherapy and the equine environment. This will provide the justification for a large-scale efficacy trial, and data for a power analysis.

PT using hippotherapy and the equine environment involves interaction between the patient and the equine. Emerging research has shown positive physiological and behavioral impacts of human-animal interactions. This PI's pilot study, which is not yet published, is the first known study to evaluate patient behavioral and physiological responses to HEI during a PT session. In Aim 3, investigators will evaluate these responses longitudinally, compare them to a control intervention, and investigate their potential moderation of patient outcomes.

Study Design A pilot, randomized-controlled trial with 24 children with NMD who will be assigned to either the PT intervention using hippotherapy and the equine environment or a standard PT control condition.

Participants Investigators will recruit 24 children from rehabilitation clinics, schools, and recreational centers around Western Montana.

Screening A research assistant will screen interested participants by phone. Those who meet initial inclusion criteria will attend a screening visit to ensure they can safely mount and dismount the equine, can provide a saliva sample, can follow simple verbal instructions, and can ambulate independently.

Sample Size The study design was determined using guidance in the NIH document Pilot Studies: Common Uses and Misuses. Investigators concluded that 80%+ power is not necessary for the current proposal because intervention efficacy is not being tested, which would require a larger sample size and length of time than this funding mechanism accommodates. Rather, the sample size is "based on practical considerations including participant flow, budgetary constraints, and the number of participants needed to reasonably evaluate goals."36 A sample size of 24 will allow sufficient participant variability to assess the feasibility of changes made to the RCT protocol and provide insight into preliminary effects of the intervention (see Preliminary Data). The investigators have assembled a strong network of recruitment partners and treatment sites (see Letters of Support) to ensure that completion of study aims with a sample of 24 subjects is achievable within the 12-month timeline.

Setting Participant baseline and post-intervention assessments and the control group treatment sessions will take place at the Pediatric Rehabilitation and Active Lifestyle (PALS) Lab at the University of Montana. The PALS lab is a 1000 ft2 space with two private assessment spaces and a waiting area for caregivers and families. The equine intervention will occur at Trotting Horse Therapeutic Riding (THTR) in Missoula, Hobby Horse Place in Polson, and Two Bear Therapeutic Riding Center in Whitefish (see Letters of Support). The facilities have accessible indoor arenas and trained therapy equines and equine professionals.

Therapists Therapists for the equine treatment are licensed physical therapists who have the recommended training to incorporate hippotherapy and the equine environment into treatment (American Hippotherapy Association (AHA) Inc. Hippotherapy Treatment Principles Part I and II). Each therapist will work with an equine professional with PATH Intl. Therapeutic Riding Instructor Certification, to ensure that therapists adhere to industry standards for safety and handling of the equines. The standard PT control intervention will be delivered by Doctor of Physical Therapy (DPT) students under the direct supervision of a licensed physical therapist.

Outcomes Assessments Pre- and post-outcomes assessments will be completed by DPT students who are trained on standardized application of all measures and under direct supervision of a licensed PT (study PI). The assessors will be blinded to subject group assignments.

Measures

The following measures will be applied to all participants:

Feasibility Fidelity Delivery of intervention Receipt of intervention Reliability: Coders for fidelity will establish ≥85% reliability by coding the same video, comparing codes, discussing any discrepancies, and reaching a consensus on any item where codes were not in agreement. This process will be repeated until the codes are congruent for ≥85% of items for sufficient reliability. Once reliability is established, the remaining videos will be divided amongst coders.

Acceptability: The engagement (PRIME-O) and enjoyment (How Happy Scale) measures described below will be used as measures of participant acceptability of the intervention.

The following measures will be collected at baseline (week 0) and post-intervention (week 9) for both groups:

GMFM-88 ABILHAND-KIDS GAS PEM-CY

The following measures will be collected at weeks 2, 4, 6, and 8 for both groups:

PRIME-O HF-HRV Salivary Oxytocin Salivary Cortisol Adaptation of How Happy Scale Behavioral Coding

Analysis Aim 1: Descriptive statistics wil be used to calculate rates of enrollment, attendance, attrition, fidelity, and outcome measure completion. Reasons for study withdrawal, missed therapy sessions, or incomplete outcome assessments will be documented. Rates will be compared between the treatment and control groups using independent samples t-tests for attendance, attrition, and measure completion and GLMMRM for fidelity.

Aim 2: Changes in outcome scores from pre- to post-intervention will be compared between groups using generalized linear mixed models for repeated measures (GLMMRM). Where available, the percent of participants who meet a minimal clinically important difference (MCID) from pre- to post-intervention will be reported.

Aim 3: HF-HRV will be calculated for the pre-, during-, and post-session intervals and compare these means. Pre-post session changes in salivary oxytocin and cortisol will be compared. HF-HRV pre-to during-session mean change and oxytocin and cortisol pre- to post-session mean changes between groups will be compared. For the behavioral data, the percentage of scans where behaviors indicate a positive or negative mood will be calculated and the average frequency of each determined and compare between groups. Longitudinal changes will be compared for all variables throughout the intervention. GLMMRM will be used for all comparisons.

ELIGIBILITY:
Inclusion Criteria:

* 1) 6-17 years old; 2) Diagnosed NMD with upper extremity impairment; 3) Able to follow simple verbal instructions in English; 4) Able to tolerate sitting on a horse continuously for 30 minutes; and 5) Meet Professional Association of Therapeutic Horsemanship International (PATH Intl.) standards for participating in mounted activities.

Exclusion Criteria:

* 1) Fear of or aversion to horses; 2) Weight over 200lbs (to protect safety and wellbeing of therapists and equines) 3) Participation in a horseback-riding program in the past 3 months; 4) Lacking independent head control; and 5) Caregivers unable to speak and read English.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
ABILHAND-KIDS | week 0 and week 9 (pre- and post-treatment)
  The ABILHAND-KIDS is a parent-report measure of a child's bimanual abilities, meaning the use of both hands, in daily activities. It asks the parent to rate their child's ability to perform 21 different bimanual daily living activities on a 3-point scale (0=impossible, 1=difficult, 2=easy).
Goal Attainment Scale (GAS) | week 0 and week 9 (pre- and post-treatment)
  The GAS is on a 5-point scale: -2, current level of performance at the time the goal is created; -1, less than expected level of performance after the 8-week intervention; 0, expected level of performance after intervention; +1, more than expected; and +2, much more than expected. Goals are determined through initial assessment and semi-structured interview with the caregiver. Goals are peer-reviewed to ensure each individual scale meets quality criteria. At the post-intervention assessment, the evaluating therapist will use direct observation and caregiver report to determine goal attainment.
Participation and Environment Measure for Children and Youth (PEM-CY) | week 0 and week 9 (pre- and post-treatment)
  A parent-report measure of child participation in activities in the home, school, and community environments, and supports or hindrances to their participation. It includes several items rated on an ordinal scale for the child's level of participation and involvement in a variety of activities. There are also short-answer questions for caregivers to elaborate on supports and barriers to their child's participation in the 3 environments, and strategies the caregivers employ to encourage/facilitate participation and involvement.
Bruininks-Oseretski Test of Motor Proficiency - Third Edition | week 0 and week 9 (pre- and post-treatment)
  The Bruininks-Oseretsky Test of Motor Proficiency - 3rd Edition is a comprehensive norm-referenced clinical measure for children and youth ages 4-21 years that covers 4 motor areas: (1) fine manual control, (2) manual coordination, (3) body coordination, and (4) strength and agility. The BOT has shown excellent test-retest reliability and good responsiveness in children with typical development and intellectual disability. Scaled scores can range from 0-20 and Standard scores can range from 0-200. Higher scores indicate better performance.
Feasibility of study protocol | 12-month study period
  We will track recruitment, screening, enrollment, retention, attendance, and outcome measure completion. We will record reasons for withdrawal, missed treatments, and incomplete outcome measures.

SECONDARY OUTCOMES:
Pediatric Rehabilitation Intervention Measure of Engagement - Observation (PRIME-O) | week 2, 4, 6, 8 during treatment period
  A 10-item observational measure of patient and service-provider engagement that accounts for affective, cognitive, and behavioral aspects of engagement. Each item is rated on a scale from 0-4.
High-Frequency Heart Rate Variability (HF-HRV) | week 2, 4, 6, 8 during treatment period
  This will be measured in the intervention group only. HF-HRV will be measured using Polar H10 heart rate sensors secured to the participant around their chest. These sensors are proven to have good reliability for measuring HF-HRV. Heart rate will be tracked for the entire therapy session in the equine environment, as well as for 5 minutes before and after the session, during which time the participant will maintain a similar level of activity, such as standing or walking, but away from the equines. For each time-interval a HF-HRV score will be assigned.
Salivary Oxytocin | week 2, 4, 6, 8 during treatment period
  Saliva will be collected from participants within 5 minutes before and after the session using the passive drool method. This is a non-invasive procedure in which the participant drools into a collection tube. Saliva samples will be stored in a medical grade freezer at the PAL lab until shipped to Salimetrics for analysis of oxytocin concentrations.
How Happy Scale | week 2, 4, 6, 8 during treatment period
  The How Happy Scale (HHS) uses a 4-point visual analog scale to evaluate a child's enjoyment of physical activity. It consists of 4 questions targeting the 4 contextual constructs of attraction, environment, social factors, and preference.
Behavioral Coding | week 2, 4, 6, 8 during treatment period
  Scan sample coding will be used to describe participant behavior during rehabilitation in the equine environment. This involves watching the treatment session and recording the behaviors of the participant at regular intervals. For this study, we will set an interval of every 1 minute, for 60 samples per session. We will record behaviors indicative of mood and engagement, such as facial expressions, positive and negative vocalizations, and engagement with therapy activities and games. We will calculate frequency of the various behaviors for each session.
Salivary Cortisol | week 2, 4, 6, 8 during treatment period
  Saliva will be collected from participants within 5 minutes before and after the session using the passive drool method. This is a non-invasive procedure in which the participant drools into a collection tube. Saliva samples will be stored in a medical grade freezer at the PAL lab until shipped to Salimetrics for analysis of oxytocin concentrations.

OTHER OUTCOMES:
Fidelity of Treatment Delivery | 4 randomly-selected treatment sessions over an 8-week period per participant
  We will measure adherence to the treatment protocol by completing a checklist of the active ingredients of the intervention that are observed in the video-recorded treatment session. The outcome will be the percentage of checklist items marked as observed.
Fidelity of Treatment Receipt | 4 randomly-selected treatment sessions over an 8-week period per participant
  The videos will be coded in Datavyu to identify participant behavior that demonstrates receipt of the intervention. Coding categories include the amount of time mounted on the horse, the amount of time completing specific participation-based activities, and completing discrete upper extremity activities such as: reaching within the base of support, reaching outside the base of support, throwing items, carrying items, holding items, grooming the horse, sweeping or mucking stalls, and clipping or latching items or doors. Each activity will be coded with information on the upper extremity(ies) being used, the type of activity occurring, and whether the activity practiced participation.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Montana, Missoula, Montana, United States

IPD SHARING:
Plan to Share IPD: No
At this time, there is no plan to share the IPD for further analysis by other researchers. We don't feel it is necessary for replicating results, as this is still a preliminary study.

REFERENCES:
- [Background] Mazzarella J, Heathcock JC. A Randomized Feasibility Study of Rehabilitation Targeting Upper Extremity Function and Participation Using Hippotherapy and the Equine Environment for Children with Cerebral Palsy and Autism Spectrum Disorder. J Integr Complement Med. 2025 Feb;31(2):196-208. doi: 10.1089/jicm.2024.0292. Epub 2024 Nov 8. PMID 39515374
- See also: PI Website — https://palslabmt.my.canva.site/umpt